CLINICAL TRIAL: NCT00636675
Title: Outcomes of Nursing Management Practice in Nursing Homes
Brief Title: CONNECT for Quality: A Study to Reduce Falls in Nursing Homes
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Carolinas Center for Medical Excellence (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00018745; 5R01NR003178 (NIH); 2R56NR003178-09 (NIH)
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Accidental Falls
Keywords: Accidental falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fall QI (Experimental): Falls QI includes quality improvement training about falls to be implement by indigenous nursing home staff with support of study personnel.
  Interventions: Behavioral: Falls QI
- Connect & Falls QI (Experimental): Connect is delivered, followed by Falls. Behavioral intervention to improve staff interaction for better care planning and execution. Connect will be delivered, followed by the Falls quality improvement intervention.
  Interventions: Behavioral: Connect

INTERVENTIONS:
Behavioral: Falls QI — Falls uses the Falls Management Program (AHRQ); it is familiar to nursing homes, uses minimal researcher time, is adaptable, and simulates real word quality improvement practices. Falls is delivered over 3 months. Components include:
  1. In-House Falls Coordinator training on content and falls processes.
  2. Case-based modules about fall prevention and tailored for various team members.
  3. Academic Detailing in which researcher consults with staff regarding challenging residents with falls.
  4. Audit and Feedback. Discussions about comparison of nursing home's current practice on fall-related process and outcome measures, and how it compares with the median and the 90th percentile of peer NHs.
  5. Toolbox: Handbook of useful measures and worksheets.
  Arms: Fall QI
Behavioral: Connect — Connect, delivered over 12 weeks, helps nursing home staff learn interactions that increase exchange of new information, number and quality of connections among staff, and improve problem-solving about patient care. Protocols:
  1. In-class learning sessions introduce interaction strategies.
  2. Relationship map protocols assist staff to examine existing interaction patterns and agree on goals for improvement. Individuals develop their own relationship maps and use them to practice new horizontal and vertical connections and self-monitoring their own interactions.
  3. Researcher facilitates authentic learning which occurs when learners directly and independently apply concepts. In-house staff volunteers and are facilitated to assume a mentoring role.
  Arms: Connect & Falls QI

SUMMARY:
Clinical trials have identified interventions that reduce adverse outcomes such as falls in nursing home (NH) residents but attempts to translate these into practice quality improvement (QI) techniques have not been successful. Using a complexity science framework, our previous study showed that low connection, information flow, and cognitive diversity among NH staff explains quality of care for complex problems such as falls. Our pilot of "Connect," a multi-component intervention that encourages staff to engage in network-building and use simple strategies to make new connections with others, enhance information flow, and use cognitive diversity, suggests that staff can improve the density and quality of their interactions. This 5-year study uses a prospective, cluster-randomized, outcome assessment blinded design, with NHs (n=16) randomized to either Connect and a falls QI program (Connect + Falls) or QI alone (Falls). About 800 residents and 576 staff will participate. Specific aims are to, in nursing homes: 1) Compare the impact of the Connect intervention plus a falls reduction QI intervention (Connect+Falls) to a falls reduction QI intervention (Falls) on fall risk reduction indicators (orthostatic blood pressure, sensory impairment, footwear appropriateness, gait; assistive device; toileting needs, environment, and psychotropic medication); 2) Compare the impact of Connect+Falls to Falls alone on fall rates and injurious falls, and determine whether these are mediated by the change in fall risk reduction indicators; 3) Compare the impact of Connect+Falls to Falls alone on complexity science measures (communication, participation in decision making, local interactions, safety climate, staff perceptions of quality) and determine whether these mediate the impact on fall risk reduction indicators and fall rates and injurious falls. Cross-sectional observations of complexity science measures are taken at baseline, at 3 months, at 6 months, and at 9 months. Resident fall risk reduction indicators, fall rates, and injurious falls are measured for the 6 months prior to the first intervention and the 6 months after the final intervention is completed. Analysis will use a 3-level mixed model to account for the complex nesting of patients and staff within nursing homes, and to control for covariates associated with fall risk, including baseline facility fall rates and staff turnover rates.

DETAILED DESCRIPTION:
Although clinical trials have identified interventions that reduce adverse outcomes such as falls in nursing home (NH) residents, attempts to translate those interventions into practice using current standard of care quality improvement (QI) programs[1, 2] have not led to expected improvements.[3, 4] Barriers encountered in previous studies point directly to a need for effective nursing management practices (NMPs).[1, 3, 5] Many studies now show that relationship-oriented NMPs such as open communication, participation in decision-making, teamwork, and leadership result in better resident outcomes.[5-10] Our recent case-studies described how NMPs work in day-to-day practice, and identified new NMPs associated with better NH care. We found that staff at all levels engaged in these NMPs, albeit erratically, suggesting that NHs have substantial untapped capacity to provide better resident care.[11-15] Thus a new intervention that fosters systematic use of NMPs may provide a foundation for more effective QI programs.

QI programs are the current standard for improving resident outcomes for common and costly conditions such as falls, pressure ulcers, pain, and depression. Such geriatric syndromes are inherently multifactorial, requiring modification of multiple risk factors to improve outcomes.[16, 17] Clinical trials using study staff to implement multiple risk factor reduction have improved resident outcomes,[18-20] but QI programs teaching existing NH staff to implement multiple risk factor reduction have not shown significant effects.[1, 21-24] One proposed reason for this failure is that QI programs seek to change individual clinician behavior but fail to account for the interactive dynamics of care. We propose that CONNECT, an intervention to foster systematic use of NMPs, will enhance the effectiveness of a Falls QI program in NHs by strengthening the one-on-one staff interactions that are necessary for clinical problem-solving about geriatric syndromes.

We have developed the Connect intervention based on complexity science and empirical research[25] to target these local interactions among staff in a new approach to facilitating organizational learning. Connect is a multicomponent intervention that includes: 1) helping staff learn new strategies to improve the effectiveness of day-to-day interactions; 2) helping staff identify important relationships and encouraging interaction at the point of care; and 3) mentoring to reinforce and sustain newly acquired interaction behaviors. Complexity science and empirical research suggest that interaction patterns determine information flow, ease of knowledge transfer, and capacity to monitor behaviors and outcomes in health care settings. [10, 26-28] Thus, Connect has the potential to improve resident outcomes when combined with QI programs for clinical problems such as falls. Falls is an excellent outcome for this initial test of Connect because: 1) there is ample evidence that multifactorial risk factor reduction interventions effectively reduce fall rates in NHs; 2) accepted practice guidelines and fall prevention programs exist;[29-32] and 3) falls is an important clinical problem in its own right.

The specific aims of this longitudinal, two arm, randomized intervention study are:

Aim 1: Compare the impact of the Connect intervention plus a falls reduction QI intervention (Connect+Falls) to the falls reduction QI intervention alone (Falls) on fall-related process measures in nursing home residents.

Aim 2 (exploratory): Compare the impact of Connect+Falls to Falls alone on fall-related outcome measures in nursing home residents, and determine whether these are mediated by the change in fall-related process measures.

Aim 3 (exploratory): Compare the impact of Connect+Falls to Falls alone on staff interaction measures as reported by NH staff, and determine whether these mediate the impact on fall-related process measures and fall-related outcome measures.

With its focus on improving local interaction, Connect is an innovative new approach targeting the learning environment to maximize NH staff's ability to adopt content learned in a Falls QI program and integrate it into knowledge and action. Our pilot work shows Connect to be feasible, acceptable and appropriate. Connect results from empirical findings; local interaction behaviors already exist in NHs, albeit to a limited extent and not in a way that effectively enables the staff to adopt evidence-based current practice for falls prevention inherent in the Falls approach. We are confident that in most NHs the capacity exists to develop and focus these behaviors using existing staff and resources and, therefore, the Connect intervention has the potential to enhance the effectiveness of Falls by promoting its adoption. Also, being a system intervention, Connect can be applied in future projects to examine the adoption of evidence-based practices for a wide variety of clinical problems such as pressure ulcers, pain, and depression. This study offers a unique opportunity to understand the circumstances in which such proven interventions (e.g., Falls) are likely to be translated into practice. Our future work will build on this study to establish correlates of the sustainability of the intervention in NHs and examine transferability to other clinical problems and other health care settings. The results of this research will be of interest to NH leadership and policy makers, particularly in light of ongoing state and national initiatives to improve care in NHs.

ELIGIBILITY:
Inclusion Criteria:

* Eligible residents will be long-term care residents at least 65 years of age who have resided in the NH at least 6 months and are likely to survive at least 6 months. Residents must be potentially at risk for falls, which we define as ambulatory or transfer-independent as recorded on the Minimum Data Set.

Exclusion Criteria:

* None.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1726 (Actual)
Dates: Start 2009-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Anderson, RN, PhD, Principal Investigator — Duke University School of Nursing; Cathleen S Colon-Emeric, MD, MHSc, Principal Investigator — Duke University
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordon M, Lanham HJ, Anderson RA, McDaniel RR Jr. Implications of complex adaptive systems theory for interpreting research about health care organizations. J Eval Clin Pract. 2010 Feb;16(1):228-31. doi: 10.1111/j.1365-2753.2009.01359.x. PMID 20367840
- [Background] McDaniel RR Jr, Lanham HJ, Anderson RA. Implications of complex adaptive systems theory for the design of research on health care organizations. Health Care Manage Rev. 2009 Apr-Jun;34(2):191-9. doi: 10.1097/HMR.0b013e31819c8b38. PMID 19322050
- [Background] Colon-Emeric CS, McConnell E, Pinheiro SO, Corazzini K, Porter K, Earp KM, Landerman L, Beales J, Lipscomb J, Hancock K, Anderson RA. CONNECT for better fall prevention in nursing homes: results from a pilot intervention study. J Am Geriatr Soc. 2013 Dec;61(12):2150-2159. doi: 10.1111/jgs.12550. Epub 2013 Nov 26. PMID 24279686
- [Background] Anderson RA, Toles MP, Corazzini K, McDaniel RR, Colon-Emeric C. Local interaction strategies and capacity for better care in nursing homes: a multiple case study. BMC Health Serv Res. 2014 Jun 5;14:244. doi: 10.1186/1472-6963-14-244. PMID 24903706
- [Background] Hall RK, Landerman LR, O'Hare AM, Anderson RA, Colon-Emeric CS. Chronic kidney disease and recurrent falls in nursing home residents: a retrospective cohort study. Geriatr Nurs. 2015 Mar-Apr;36(2):136-41. doi: 10.1016/j.gerinurse.2014.12.012. Epub 2015 Jan 20. PMID 25616732
- [Background] Marcum ZA, Gurwitz JH, Colon-Emeric C, Hanlon JT. Pills and ills: methodological problems in pharmacological research. J Am Geriatr Soc. 2015 Apr;63(4):829-30. doi: 10.1111/jgs.13371. No abstract available. PMID 25900504
- [Background] Mewshaw J, Bailey DE Jr, Porter KA, Anderson AL, Anderson RA, Burd AL, Colon-Emeric C, Corazzini KN. A novel program for ABSN students to generate interest in geriatrics and geriatric nursing research. J Nurs Educ Pract. 2017 Jun;7(6):95-99. doi: 10.5430/jnep.v7n6p95. Epub 2017 Feb 5. PMID 28435479
- [Result] Utley-Smith Q, Colon-Emeric CS, Lekan-Rutledge D, Ammarell N, Bailey D, Corazzini K, Piven ML, Anderson RA. The Nature of Staff - Family Interactions in Nursing Homes: Staff Perceptions. J Aging Stud. 2009 Aug;23(3):168-177. doi: 10.1016/j.jaging.2007.11.003. PMID 19649311
- [Result] Colon-Emeric CS, Lekan D, Utley-Smith Q, Ammarell N, Bailey D, Corazzini K, Piven ML, Anderson RA. Barriers to and facilitators of clinical practice guideline use in nursing homes. J Am Geriatr Soc. 2007 Sep;55(9):1404-9. doi: 10.1111/j.1532-5415.2007.01297.x. PMID 17767682
- [Result] Piven ML, Ammarell N, Lekan-Rutledge D, Utley-Smith Q, Corazzini KN, Colon-Emeric CS, Bailey D, Anderson RA. Paying attention: A leap toward quality care. Director. 2007 Winter;15(1):58-60, 62-3. No abstract available. PMID 17710200
- [Result] Corazzini KN, Lekan-Rutledge D, Utley-Smith Q, Piven ML, Colon-Emeric CS, Bailey D, Ammarell N, Anderson RA. "The Golden Rule": Only a starting point for quality care. Director. 2005;14(1):255-293. PMID 17334452
- [Result] Utley-Smith Q, Bailey D, Ammarell N, Corazzini K, Colon-Emeric CS, Lekan-Rutledge D, Piven ML, Anderson RA. Exit interview-consultation for research validation and dissemination. West J Nurs Res. 2006 Dec;28(8):955-73. doi: 10.1177/0193945905282301. PMID 17099107
- [Result] Piven ML, Ammarell N, Bailey D, Corazzini K, Colon-Emeric CS, Lekan-Rutledge D, Utley-Smith Q, Anderson RA. MDS coordinator relationships and nursing home care processes. West J Nurs Res. 2006 Apr;28(3):294-309. doi: 10.1177/0193945905284710. PMID 16585806
- [Result] Colon-Emeric CS, Ammarell N, Bailey D, Corazzini K, Lekan-Rutledge D, Piven ML, Utley-Smith Q, Anderson RA. Patterns of medical and nursing staff communication in nursing homes: implications and insights from complexity science. Qual Health Res. 2006 Feb;16(2):173-88. doi: 10.1177/1049732305284734. PMID 16394208
- [Result] Anderson RA, Ammarell N, Bailey D Jr, Colon-Emeric C, Corazzini KN, Lillie M, Piven ML, Utley-Smith Q, McDaniel RR Jr. Nurse assistant mental models, sensemaking, care actions, and consequences for nursing home residents. Qual Health Res. 2005 Oct;15(8):1006-21. doi: 10.1177/1049732305280773. PMID 16221876
- [Result] Anderson RA, Ammarell N, Bailey DE, Colon-Emeric C, Corazzini K, Lekan-Rutledge D, Piven ML, Utley-Smith Q. The power of relationship for high-quality long-term care. J Nurs Care Qual. 2005 Apr-Jun;20(2):103-6. doi: 10.1097/00001786-200504000-00003. No abstract available. PMID 15839289
- [Result] Anderson RA, Crabtree BF, Steele DJ, McDaniel RR Jr. Case study research: the view from complexity science. Qual Health Res. 2005 May;15(5):669-85. doi: 10.1177/1049732305275208. PMID 15802542
- [Result] Colon-Emeric CS, Plowman D, Bailey D, Corazzini K, Utley-Smith Q, Ammarell N, Toles M, Anderson R. Regulation and mindful resident care in nursing homes. Qual Health Res. 2010 Sep;20(9):1283-94. doi: 10.1177/1049732310369337. Epub 2010 May 17. PMID 20479137
- [Result] Toles M, Anderson RA. State of the science: relationship-oriented management practices in nursing homes. Nurs Outlook. 2011 Jul-Aug;59(4):221-7. doi: 10.1016/j.outlook.2011.05.001. PMID 21757079
- [Result] Colon-Emeric CS, Pinheiro SO, Anderson RA, Porter K, McConnell E, Corazzini K, Hancock K, Lipscomb J, Beales J, Simpson KM. Connecting the learners: improving uptake of a nursing home educational program by focusing on staff interactions. Gerontologist. 2014 Jun;54(3):446-59. doi: 10.1093/geront/gnt043. Epub 2013 May 23. PMID 23704219
- [Result] Ausserhofer D, Anderson RA, Colon-Emeric C, Schwendimann R. First evidence on the validity and reliability of the Safety Organizing Scale-Nursing Home version (SOS-NH). J Am Med Dir Assoc. 2013 Aug;14(8):616-22. doi: 10.1016/j.jamda.2013.03.016. Epub 2013 May 14. PMID 23684122
- [Result] Simpson KM, Porter K, McConnell ES, Colon-Emeric C, Daily KA, Stalzer A, Anderson RA. Tool for evaluating research implementation challenges: a sense-making protocol for addressing implementation challenges in complex research settings. Implement Sci. 2013 Jan 2;8:2. doi: 10.1186/1748-5908-8-2. PMID 23281623
- [Result] Anderson RA, Corazzini K, Porter K, Daily K, McDaniel RR Jr, Colon-Emeric C. CONNECT for quality: protocol of a cluster randomized controlled trial to improve fall prevention in nursing homes. Implement Sci. 2012 Feb 29;7:11. doi: 10.1186/1748-5908-7-11. PMID 22376375
- [Result] Colon-Emeric C, Toles M, Cary MP Jr, Batchelor-Murphy M, Yap T, Song Y, Hall R, Anderson A, Burd A, Anderson RA. Sustaining complex interventions in long-term care: a qualitative study of direct care staff and managers. Implement Sci. 2016 Jul 16;11:94. doi: 10.1186/s13012-016-0454-y. PMID 27422011
- [Result] Colon-Emeric CS, Corazzini K, McConnell E, Pan W, Toles M, Hall R, Batchelor-Murphy M, Yap TL, Anderson AL, Burd A, Anderson RA. Study of Individualization and Bias in Nursing Home Fall Prevention Practices. J Am Geriatr Soc. 2017 Apr;65(4):815-821. doi: 10.1111/jgs.14675. Epub 2017 Feb 10. PMID 28186618
- [Derived] Colon-Emeric CS, Corazzini K, McConnell ES, Pan W, Toles M, Hall R, Cary MP Jr, Batchelor-Murphy M, Yap T, Anderson AL, Burd A, Amarasekara S, Anderson RA. Effect of Promoting High-Quality Staff Interactions on Fall Prevention in Nursing Homes: A Cluster-Randomized Trial. JAMA Intern Med. 2017 Nov 1;177(11):1634-1641. doi: 10.1001/jamainternmed.2017.5073. PMID 28973516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We invited 69 nursing homes (NHs) with > 89 beds participating in Medicare and Medicaid within 100 miles of Duke, and included the first 24 homes responding. Staff were invited as part of their facility's quality improvement (QI) initiatives. We used a random sample of 50 residents from each facility for chart abstraction.
Groups:
- Fall QI: Falls QI includes quality improvement training about falls to be implement by indigenous nursing home staff with support of study personnel.
  Falls QI: Falls uses the Falls Management Program (AHRQ); it is familiar to nursing homes, uses minimal researcher time, is adaptable, and simulates real word quality improvement practices. Falls is delivered over 3 months. Components include:
  1. In-House Falls Coordinator training on content and falls processes.
  2. Case-based modules about fall prevention and tailored for various team members.
  3. Academic Detailing in which researcher consults with staff regarding challenging residents with falls.
  4. Audit and Feedback. Discussions about comparison of nursing home's current practice on fall-related process and outcome measures, and how it compares with the median and the 90th percentile of peer NHs.
  5. Toolbox: Handbook of useful measures and worksheets.
- Connect & Falls QI: Connect is delivered, followed by Falls. Behavioral intervention to improve staff interaction for better care planning and execution. Connect will be delivered, followed by the Falls quality improvement intervention.
  Connect: Connect, delivered over 12 weeks, helps nursing home staff learn interactions that increase exchange of new information, number and quality of connections among staff, and improve problem-solving about patient care. Protocols:
  1. In-class learning sessions introduce interaction strategies.
  2. Relationship map protocols assist staff to examine existing interaction patterns and agree on goals for improvement. Individuals develop their own relationship maps and use them to practice new horizontal and vertical connections and self-monitoring their own interactions.
  3. Researcher facilitates authentic learning which occurs when learners directly and independently apply concepts. In-house staff volunteers and are facilitated to assume a mentoring role.
Period: Overall Study
Arm/Group | Fall QI | Connect & Falls QI
Started | 951 | 775
Completed | 811 | 734
Not Completed | 140 | 41
Not completed — Lost to Follow-up | 121 | 31
Not completed — Withdrawal by Subject | 19 | 10

BASELINE CHARACTERISTICS:
Population: Participants who completed all follow up measures.
Groups:
- Falls Qualty Improvement (QI): Falls QI includes quality improvement training about falls to be implement by indigenous nursing home staff with support of study personnel.
  Falls QI: Falls uses the Falls Management Program; it is familiar to nursing homes, uses minimal researcher time, is adaptable, and simulates real word quality improvement practices. Falls is delivered over 3 months. Components include:
  1. In-House Falls Coordinator training on content and falls processes.
  2. Case-based modules about fall prevention and tailored for various team members.
  3. Academic Detailing in which researcher consults with staff regarding challenging residents with falls.
  4. Audit and Feedback. Discussions about comparison of nursing home's current practice on fall-related process and outcome measures, and how it compares with the median and the 90th percentile of peer NHs.
  5. Toolbox: Handbook of useful measures and worksheets.
- Connect & Falls Quality Improviement (QI): Connect is delivered, followed by Falls. Behavioral intervention to improve staff interaction for better care planning and execution. Connect will be delivered, followed by the Falls quality improvement intervention.
  Connect: Connect, delivered over 12 weeks, helps nursing home staff learn interactions that increase exchange of new information, number and quality of connections among staff, and improve problem-solving about patient care. Protocols:
  1. In-class learning sessions introduce interaction strategies.
  2. Relationship map protocols assist staff to examine existing interaction patterns and agree on goals for improvement. Individuals develop their own relationship maps and use them to practice new horizontal and vertical connections and self-monitoring their own interactions.
  3. Researcher facilitates authentic learning which occurs when learners directly and independently apply concepts. In-house staff volunteers and are facilitated to assume a mentoring role.
- Total: Total of all reporting groups
Arm/Group | Falls Qualty Improvement (QI) | Connect & Falls Quality Improviement (QI) | Total
Number analyzed (Participants) | 743 | 658 | 1401
Age, Categorical [Count of Participants; unit: Participants] — Population: Not all participants completed the surveys and/or they did not complete all items and so the baseline numbers differ from the participant flow chart
  Participants
    Age: number analyzed (Participants) | 731 | 646 | 1377
    Age: <=18 years | 0 | 0 | 0
    Age: Between 18 and 65 years | 615 | 509 | 1124
    Age: >=65 years | 116 | 137 | 253
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all participants completed the surveys and/or they did not complete all items and so the baseline numbers differ from the participant flow chart
  Participants
    number analyzed (Participants) | 706 | 626 | 1332
    Female | 600 | 554 | 1154
    Male | 106 | 72 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 34
  Not Hispanic or Latino | 681 | 599 | 1280
  Unknown or Not Reported | 49 | 38 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 21 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 337 | 281 | 618
  White | 316 | 296 | 612
  More than one race | 11 | 14 | 25
  Unknown or Not Reported | 57 | 51 | 108
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 743 | 658 | 1401

OUTCOME MEASURES:

1. Primary Outcome: Fall Related Process Measures
Description: Mean of the total number of fall risk reduction indicators (steps staff have taken to reduce fall risk) that were documented in residents with high fall risk. These included orthostatic blood pressure measurement/intervention; sensory impairment evaluation/intervention; footwear; exercise/assistive device intervention; toileting schedule; environmental modification; psychoactive medication reduction; and vitamin D supplements. Note that this measure is NOT related to staff but rather residents in the nursing home, therefore the numbers are different from participant flow. The residents were not considered enrolled participants in the study.
Time Frame: 6 months post intervention
Population: Residents with prior fall
Measure: Mean (Standard Deviation); unit: number of fall risk reduction indicators
Arm/Group | Fall QI | Connect & Falls QI
Number analyzed (Participants) | 907 | 887
number of fall risk reduction indicators | 3.3 (1.6) | 3.2 (1.5)

2. Secondary Outcome: Fall Rates
Description: Numerator: number of falls occurring in a 6 month period, denominator: number of bed days for resident. Rate adjusted for baseline rate and casemix. Note that this measure is NOT related to staff but rather residents in the nursing home. The residents were not considered enrolled participants in the study.
Time Frame: 6 months post intervention
Population: Residents with at least one prior fall
Measure: Median (Inter-Quartile Range); unit: fall rate
Arm/Group | Fall QI | Connect & Falls QI
Number analyzed (Participants) | 907 | 887
fall rate | 4.06 [2.04 to 8.11] | 4.06 [2.03 to 8.11]

3. Secondary Outcome: Change in Weighted Average of Staff Interaction Scales
Description: This is a summary measure of 7 staff surveys using the weighted average on a 1-5 Likert scale with 5 indicating the highest (best) quality. Scales include Communication Openness, Accuracy, and Timeliness; Participation in Decision Making, Local Interaction Strategies, Safety Climate, and Staff Perceptions of Quality. Number presented is the change from baseline attributable to the intervention. Higher numbers represent a greater change attributable to the intervention.
Time Frame: baseline to post intervention, an average of 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fall QI | Connect & Falls QI
Number analyzed (Participants) | 743 | 658
units on a scale | NA (NA) — The CONNECT intervention was not delivered to this group, therefore no change attributable to intervention was calculated. | .03 (0.02)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events for participating staff
Arm/Group | Fall QI | Connect & Falls QI
All-Cause Mortality (participants affected / at risk) | 0/811 | 0/734
Serious Adverse Events (participants affected / at risk) | 0/811 | 0/734
Other Adverse Events (participants affected / at risk) | 0/811 | 0/734

LIMITATIONS AND CAVEATS:
While randomized, the relatively small number of nursing homes (N = 24) likely resulted in imbalances in facility, staff, and resident-level factors by chance alone. We were limited to one geographic region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No